CLINICAL TRIAL: NCT02976155
Title: The Effect of a Standard Enteral Nutrition Protocol on Critically Ill Patients: a Multiple-center, Prospective, Before-after Study
Brief Title: The Effect of Standardized Enteral Nutrition on Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Department of Emergency Medicine, People's Hospital of Shaoxing, Shaoxing, China. (Unknown); Department of Emergency Medicine, Wenzhou Central Hospital, Wenzhou, China. (Unknown); Department of Emergency Medicine, The First People's Hospital of Hangzhou, Hangzhou, China. (Unknown); Department of Emergency Medicine, The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, China. (Unknown); Sir Run Run Shaw Hospital (Other); Emergency Department, The First People's Hospital of Huzhou, Huzhou, China. (Unknown); Department of Critical Care Medicine, The First People's Hospital of Xiaoshan District, Hangzhou, China. (Unknown); Emergency Department, Jinhua Hospital of Zhejiang University, Jinhua, China. (Unknown); Department of Critical Care Medicine, The First People's Hospital of Fuyang district, Hangzhou, China. (Unknown); Department of Critical Care Medicine, Beilun District People's Hospital, Ningbo, China. (Unknown); The Affiliated Hospital of Hangzhou Normal University (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); Yuyao People's Hospital (Other); Department of Emergency Intensive Care Unit, The Second Hospital of Jiaxing, No 1518, Huanchengbei Rd, Jiaxing, China. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 87783921
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2018-09

CONDITIONS: Critically Ill
Keywords: critically ill, intensive care, enteral nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Before-after study model
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-intervention (No Intervention): enteral nutrition according routine practice
- Post-intervention (Experimental): The intervention in this arm is the application of a standard enteral nutrition protocol
  Interventions: Other: A standard enteral nutrition protocol

INTERVENTIONS:
Other: A standard enteral nutrition protocol — Patients in the experimental arm, the practice of enteral nutrition will based on a standard protocol. The core content of this protocol includes five step：1. Whether the participants need nutrition therapy? 2. The choice of nutrition way? 3. Nasogastric tube or nasointestinal tube? 4. The choice of enteral nutrition type? 5. The target calorie and protein of the participants? And how to achieve these target？(In this study, the practice of the above protocol is the only intervention).
  Arms: Post-intervention

SUMMARY:
The goal of this study is to evaluate whether a standard enteral nutrition protocol can improve the efficiency in achieving nutritional goals and improve prognosis in critically ill patients.

DETAILED DESCRIPTION:
As investigators all know, the nutrition status in critically ill patients is associated with the prognosis of these patients. And it has been confirmed that early enteral nutrition results in better outcome. However,some epidemiological investigation reported that in most intensive care unit, the phenomenon of delayed feeding or under feeding are not uncommon. In 2007, a study reported that the percentage of early enteral nutrition within 48h is 64%, based on mechanical ventilated patients in 208 intensive care unit nationally. Other study indicated that the calorie supported by the enteral nutrition only constitute 50% of the target calorie. Several studies have showed that the application of a standard enteral nutrition protocol could result in an improvement in the delivery of enteral feedings to patients. However, there is no such study in China.The goal of this study is to evaluate whether a standard enteral nutrition protocol can improve the efficiency in achieving nutritional goals and improve prognosis in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients who is expected the length of ICU stay for more than 3 days

Exclusion Criteria:

* Patients who can obtain enough calorie through independent oral feeding. Patients aged less than 18 years. Patients who are pregnant or breastfeeding. Patients who are burned. Patients with malignant tumor terminal stages of diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients receiving enteral nutrition in patients receiving any type of nutrition | 7 days after ICU admission
The time from hospital admission to the begain Enteral nutrition. | 7 days after ICU admission
The time from hospital admission to achieve the target calorie. | 7 days after ICU admission
The proportion of patients receiving parenteral nutrition in patients receiving any type of nutrition | 7 days after ICU admission
The proportion of patients receiving Enteral plus supplement parenteral in patients receiving any type of nutrition | 7 days after ICU admission

SECONDARY OUTCOMES:
ICU mortality. | From date of the ICU admission until discharge form ICU,assessed up to 12 months
Hospital mortality. | From date of the ICU admission until discharge form hospital,assessed up to 12 months
ICU length of stay | From date of the ICU admission until discharge form ICU,assessed up to 12 months
Duration of mechanical ventilation. | From date of the initiation of mechanical ventilation until weaning,assessed up to 12 months
ICU fee. | From date of the ICU admission until discharge form ICU,assessed up to 12 months
The incidence of complications(Diarrhea , abdominal distension, nausea and vomiting.) | From date of the ICU admission until discharge form ICU,assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang university, school of medicine., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang L, Huang X, Wu C, Tang J, Li Q, Feng X, He T, Wang Z, Gao J, Ruan Z, Hong W, Lai D, Zhao F, Huang Z, Lu Z, Tang W, Zhu L, Zhang B, Wang Z, Shen X, Lai J, Ji Z, Fu K, Hong Y, Dai J, Hong G, Xu W, Wang Y, Xie Y, Chen Y, Zhu X, Ding G, Gu L, Zhang M. The effects of an enteral nutrition feeding protocol on critically ill patients: A prospective multi-center, before-after study. J Crit Care. 2020 Apr;56:249-256. doi: 10.1016/j.jcrc.2020.01.018. Epub 2020 Jan 17. PMID 31986368